CLINICAL TRIAL: NCT03655249
Title: Effects of Autogenic Drainage on Ventilation Inhomogeneity in Patients With Cystic Fibrosis
Brief Title: Effects of AD on VI in Patients With CF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018/22FEV/079
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Cystic Fibrosis
Keywords: Multiple breath washout; Electrical impedance tomography; Lung clearance index; Chest physiotherapy; Autogenic drainage; Cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Participants receive one of two interventions during the first day, and receive the alternative intervention the following day.
  Interventions are : aerosoltherapy + autogenic drainage or aerosoltherapy alone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asl + CPT (Experimental): Aerosotherapy + Autogenic drainage
  Interventions: Other: Autogenic drainage; Drug: Aerosoltherapy
- Asl (Active Comparator): Aerosoltherapy alone
  Interventions: Drug: Aerosoltherapy

INTERVENTIONS:
Other: Autogenic drainage — Autogenic drainage is an airway clearance technique that attempts to obtain the optimal airflow to evacuate the secretions. This technique uses modulation of inspiratory and expiratory airflow at different breathing level within the vital capacity.
  Arms: Asl + CPT
Drug: Aerosoltherapy — Aerosolized drugs are individualized for each participants, in line with current standardized practice in our hospital. Those drugs will not be modified for the purpose of this study.

SUMMARY:
This study will investigate the effects of a chest physiotherapy manual technique (autogenic drainage) on ventilation inhomogeneity in patients with cystic fibrosis. Lung clearance index (LCI) is the primary outcome

DETAILED DESCRIPTION:
This is a cross-over intervention assessing the effect of autogenic drainage on ventilation inhomogeneity in patients with cystic fibrosis.

Electrical impedance tomography and multiple breath nitrogen washout will be performed before, immediatly after and 2h post intervention. Each participant will receive either aerosoltherapy alone or in combination with chest physiotherapy on 2 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis diagnosis
* FEV1 > 40%
* Able to sustain 30min of chest physiotherapy

Exclusion Criteria:

* Presence of Burkoldheria cepacia or non tuberculous mycobacteria
* Orthopedic, neuromuscular or cardiac disorder likely to impact respiratory system
* Need for supplemental oxygen
* Cardiac pacemaker or internal cardiac defibrillator

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Lung Clearance Index | Up to 2 weeks
  LCI will be measured before, immediately after and 2h after the experimental or control conditions as well as before and after an hospitalization.

SECONDARY OUTCOMES:
Impedance variation | Up to 1 hour
  Impedance change in different lung zones

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reychler, PT, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium